CLINICAL TRIAL: NCT07088263
Title: A Prospective, Multicenter Phase Ⅲ Clinical Trial of Adaptive Chemotherapy for Advanced Breast Cancer After Standard Treatment
Brief Title: Adaptive Chemotherapy for the Treatment of Advanced Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-081
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Vinorelbine; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemotherapy repeated every 28 days (Experimental): Chemotherapy regimens, including gemcitabine, vinorelbine, eribulin, or utidelone.
  Gemcitabine 1000 mg/m², IV, days 1, 8; or Vinorelbine 25 mg/m², IV, days 1, 8; Vinorelbine 60-80 mg/m², Po., days 1, 8; Eribulin 1.4 mg/m², IV, days 1, 8; Utidelone 30 mg/m², IV, days 1-5; All cycles repeated every 28 days.
  Interventions: Drug: Gemcitabine, Vinorelbine, Eribulin, or Utidelone
- Chemotherapy repeated every 21 days (Active Comparator): Chemotherapy regimens, including gemcitabine, vinorelbine, eribulin, or utidelone.
  Gemcitabine 1000 mg/m², IV, days 1, 8; or Vinorelbine 25 mg/m², IV, days 1, 8; Vinorelbine 60-80 mg/m², Po., days 1, 8; Eribulin 1.4 mg/m², IV, days 1, 8; Utidelone 30 mg/m², IV, days 1-5; All cycles repeated every 21 days.
  Interventions: Drug: Gemcitabine, Vinorelbine, Eribulin, or Utidelone

INTERVENTIONS:
Drug: Gemcitabine, Vinorelbine, Eribulin, or Utidelone — Gemcitabine, Vinorelbine, Eribulin, or Utidelone is recieved every 28 days. The chemotherapy interval is one cycle every 28 days.

SUMMARY:
The primary objective of this study is to explore the efficacy and safety of adaptive therapy in the treatment of advanced breast cancer progressive after standard treatment.

DETAILED DESCRIPTION:
This is a prospective, multicenter phase Ⅲ clinical Trial. The objective of the study is to evaluate the efficacy and safety of adaptive chemotherapy vs. conventional chemotherapy in the treatment of advanced breast cancer progressive after standard treatment. The therapy regimen, primarily including gemcitabine, vinorelbine, or eribulin, will be selected by the investigator based on current guidelines, available treatments, and an assessment of the patient's clinical status, preferences, and financial situation. This study is designed to recruit up to 192 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Understands and voluntarily signs the informed consent form.
* ECOG PS of 0 or 1.
* Expected survival: >3 months
* Histologically or cytologically confirmed advanced invasive breast cancer.
* Histological type: HR+/HER2- or HR-/HER2-. HR positivity is defined as ER and/or PR expression in ≥1% of tumor cells by IHC. HER2 negativity is defined according to the ASCO-CAP HER2 guidelines: IHC intensity of 0 or 1+, or IHC intensity of 2+ with negative in situ hybridization results.
* Previous failure of first-line treatment for metastatic disease. For HR+/HER2- patients: at least received endocrine therapy combined with CDK4/6 inhibitors. TNBC patients at least received chemotherapy combined with PD-1 inhibitors (if PD-L1 CPS ≥1), or PARP inhibitor treatment (if germline BRCA mutations), except for TNBC patients with known germline BRCA mutations whom the attending physician deems them unable or unsuitable for PARP inhibitor treatment.
* At least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Adequate organ function including bone marrow, renal function, hepatic function, and cardiac reserve.
* Premenopausal women must use medically acceptable contraception during the study.
* Compliance with the study protocol.

Exclusion Criteria:

* The investigator considers that the presence of the following factors would be unfavorable to the subject's participation in the study or may affect protocol compliance, such as uncontrolled hypertension, persistent or active infection, etc.
* Persistent toxicities caused by previous anti-tumor treatment that have not improved to ≤ Grade 2 or baseline levels.
* Neoplastic spinal cord compression or active brain metastases.
* Significant third-space fluid retention (e.g., ascites or pleural effusion).
* Uncontrolled infection requiring treatment with intravenous antibiotic.
* Active or uncontrolled hepatitis B or hepatitis C virus infection.
* Uncontrolled or significant heart disease.
* Suspected ILD/non-infectious pneumonia.
* Active autoimmune disease or inflammatory disease (including inflammatory bowel disease.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-07-24 (Estimated); Study Completion 2028-06-24 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 12 months
  progression-free survival (PFS): The interval time from the date of initiation treatment after recruit to the date of the first documented disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No